CLINICAL TRIAL: NCT00637247
Title: A Phase 2 Randomized, Double-Blind, Multicenter Trial of Amplimexon® Plus Gemcitabine Versus Gemcitabine Plus Placebo in Patients With Metastatic Chemotherapy Naïve Pancreatic Adenocarcinoma (Stage IV)
Brief Title: A Randomized Study of Amplimexon (Imexon) With Gemcitabine in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AmpliMed Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMP-019
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Neoplasms
Keywords: pancreatic cancer; metastatic; chemotherapy naive
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — 4-imino-1,3-diazabicyclo(3.1.0)hexan-2-one; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- imexon + gemcitabine (Experimental): imexon + gemcitabine
  Interventions: Drug: imexon in combination with gemcitabine
- Placebo + gemcitabine (Active Comparator): Placebo in combination with gemcitabine
  Interventions: Drug: imexon placebo + gemcitabine

INTERVENTIONS:
Drug: imexon in combination with gemcitabine — 875 mg/m^2 imexon IV + 1000 mg/m^2 gemcitabine IV
  Other Names: Amplimexon, Gemzar
  Arms: imexon + gemcitabine
Drug: imexon placebo + gemcitabine — imexon placebo IV + 1000 mg/m^2 gemcitabine IV
  Other Names: Gemzar
  Arms: Placebo + gemcitabine

SUMMARY:
The purpose of this study is to determine if imexon in combination with gemcitabine could improve overall survival as compared to gemcitabine alone in subjects with pancreatic cancer that has spread to other organs such as the liver or lungs. The study will also look at the safety of the combination as compared to gemcitabine alone. Participants in the study will be randomly assigned to either treatment and neither the participant or their doctors will know which treatment they will be receiving.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed, chemotherapy naive, metastatic pancreatic adenocarcinoma (Stage IV). This does not include patients with only locally advanced pancreatic cancer.
2. At least one unidimensional measurable metastatic lesion by contrast enhanced CT scan (or MRI in patients ineligible for contrast enhanced CT) that are outside any prior radiation port.
3. Age at least 18 years.
4. ECOG performance status 0 or 1.
5. No prior chemotherapy or radiation therapy.
6. Projected life expectancy at least 2 months.
7. If female, neither pregnant nor lactating.
8. If of child bearing potential must agree to, and be able to use adequate contraception.
9. Concomitant disease: No respiratory insufficiency requiring oxygen therapy; no angina at rest; no myocardial infarction in previous 3 months; no life threatening ventricular arrhythmias. No uncompensated CHF or NY Heart Association class 3 or 4 cardiac disease.
10. No other concurrent active malignancy.
11. No infection requiring parenteral antibiotic therapy at the start of protocol treatment.
12. Laboratory values within the following criteria:

    Hgb greater than or equal to 9 gm/dL WBC greater than or equal 3,500/mm^3 ANC greater than or equal 1,500/mm^3 Platelet count greater than or equal 100,000/mm^3 Creatinine greater than or equal 2.0 Bilirubin less than or equal to 2.0 Hepatic enzymes (AST, ALT) less than or equal 3 times upper limit of normal (ULN)
13. G6PD level greater than or equal lower limit of normal (LLN).
14. Able to render informed consent and follow protocol requirements.

Exclusion Criteria:

1. Patients with locally advanced, non-metastatic pancreas cancer (Stage III or below).
2. Age less than 18 years.
3. ECOG performance status 2 or greater.
4. Prior anticancer drug therapy for metastatic disease.
5. Ascites.
6. Prior abdominal or thoracic surgery < 4 weeks before the start of therapy.
7. Current or prior brain metastases. Brain MRI or CT required pre-registration only if the patient has CNS symptoms indicating a need for evaluation.
8. Life expectancy projected less than 2 months.
9. Pregnancy or lactation.
10. Unable or unwilling to utilize medically acceptable contraception if of childbearing potential.
11. Laboratory parameters outside of specified ranges, (see above).
12. Infection requiring parenteral antibiotics.
13. NY Heart Association stage 3 or 4 heart disease.
14. Unable to render informed consent.
15. Failure to meet any of the eligibility criteria as outlined above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Hersh, MD, Study Director — AmpliMed Corporation; Steven Cohen, MD, Principal Investigator — Fox Chase Cancer Center
Locations (48):
- United States (48):
  - Birmingham Hematology and Oncology- US Oncology, Birmingham, Alabama
  - AZ Onc Associates D.B.A. Hematology Oncology- US Oncology, Tucson, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Rocky Mountain Cancer Center- US Oncology, Denver, Colorado
  - Ocala Oncology Center- US Oncology, Ocala, Florida
  - Cancer Centers of Florida- US Oncology, Orlando, Florida
  - Peachtree Hematology and Oncology Consultants, Atlanta, Georgia
  - Hematology Oncology Associates of Illinois- US Oncology, Chicago, Illinois
  - Cancer Care & Hematolog Specialists of Chicagoland- US Oncology, Niles, Illinois
  - Central Indiana Cancer Centers- US Oncology, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Hope Center- US Oncology, Terre Haute, Indiana
  - University of Kentucky, Hematology/Oncology/BMT Clinical Research, Lexington, Kentucky
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Kansas City Cancer Center, LLC- US Oncology, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada- US Oncology, Las Vegas, Nevada
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Hematology Oncology Associates, Mount Holly, New Jersey
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - University of New Mexico Cancer Center South, Las Cruces, New Mexico
  - New Mexico Cancer Care Associates- US Oncology, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cancer Center of North Carolina- US Oncology, Raleigh, North Carolina
  - Medical Onc Assoc of Wyoming Valley, PC- US Oncology, Kingston, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Associates in Hematology-Oncology P.C. US Oncology, Upland, Pennsylvania
  - Reading Hospital Regional Medical Center, West Reading, Pennsylvania
  - Sanford Clinic, Sioux Falls, South Dakota
  - Texas Oncology - Amarillo- US Oncology, Amarillo, Texas
  - Mamie Mcfaddin Ward Cancer Center, Texas Oncology- US Oncology, Beaumont, Texas
  - Texas Oncology P.A.- Bedford- US Oncology, Bedford, Texas
  - Texas Cancer Center at Medical City- US Oncology, Dallas, Texas
  - Texas Oncology P.A. - Dallas- US Oncology, Dallas, Texas
  - Methodist Charlton Cancer Center - Texas Oncology- US Oncology, Dallas, Texas
  - Texas Oncology - Odessa- US Oncology, Odessa, Texas
  - Scott and White Hospital and Clinics, Temple, Texas
  - Texas Oncology Cancer Care and Research Center- US Oncology, Waco, Texas
  - Texoma Cancer Center- US Oncology, Wichita Falls, Texas
  - Virginia Oncology Associates- US Oncology, Norfolk, Virginia
  - Onc & Hematology Assoc. of Southern VA, Inc D.B.A. - US Oncology, Salem, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Cancer Care Northwest- US Oncology, Spokane, Washington
  - Northwest Cancer Specialists- US Oncology, Vancouver, Washington

REFERENCES:
- [Background] Cohen SJ, Zalupski MM, Conkling P, Nugent F, Ma WW, Modiano M, Pascual R, Lee FC, Wong L, Hersh E. A Phase 2 Randomized, Double-Blind, Multicenter Trial of Imexon Plus Gemcitabine Versus Gemcitabine Plus Placebo in Patients With Metastatic Chemotherapy-naive Pancreatic Adenocarcinoma. Am J Clin Oncol. 2018 Mar;41(3):230-235. doi: 10.1097/COC.0000000000000260. PMID 26709865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from April 2008 to May 2009. Enrollment occurred at 34 clinical centers in the United States.
Groups:
- Amplimexon (Imexon) + Gemcitabine: Amplimexon 875 mg/m^2 + gemcitabine 1000 mg/m^2
- Imexon Placebo + Gemcitabine: Placebo 875 mg/m^2+ gemcitabine 1000 mg/m^2
Period: Overall Study
Arm/Group | Amplimexon (Imexon) + Gemcitabine | Imexon Placebo + Gemcitabine
Started | 72 | 70
Completed | 72 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amplimexon (Imexon) + Gemcitabine | Imexon Placebo + Gemcitabine | Total
Number analyzed (Participants) | 72 | 70 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 31 | 65
  >=65 years | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (10.6) | 64.9 (11.1) | 65.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 41 | 39 | 80
Region of Enrollment [Number; unit: participants]
  United States | 72 | 70 | 142

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival for the Intent to Treat Population
Description: To compare the overall survival duration of the two treatment arms. Overall survival is measured from the time of randomization until reported death. Subjects were censored at last time known alive if lost to follow-up. Alive patients were censored at the last survival follow-up. Follow-up was monthly after off study treatment.
Time Frame: up to 2 years
Population: Intention to treat with subjects who were alive at the time of the survival analysis or lost to follow-up were considered censored at the last date the subject was known to be alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amplimexon (Imexon) + Gemcitabine | Imexon Placebo + Gemcitabine
Number analyzed (Participants) | 72 | 70
months | 5.2 [4.2 to 6.7] | 6.8 [4.9 to 8.5]
Statistical Analysis 1: Comparison: Amplimexon (Imexon) + Gemcitabine vs Imexon Placebo + Gemcitabine; The hypothesis that survival curves were equal in the two treatment groups was tested with a one-sided logrank test at the alpha-0.2 level, one sided. The power of this test is 80% for detecting the hypothesized increase in median survival of 2.4 months for subjects in the experimental arm; Test type: Superiority or Other; p = 0.2, Log Rank

2. Primary Outcome: To Evaluate and Compare the Tolerability and Toxicity of the Two Treatment Arms by Comparing Adverse Events
Description: Number of Participants with Adverse Events were compared between the two arms to detect any differences in number or types of events
Time Frame: Adverse events were collected from the time of treatment until the participant went off study treatment, an average of 4 months
Population: This includes only those subjects that received at least 1 dose of study treatment. There were 67 subjects in the imexon + gemcitabine arm and 68 in the placebo + gemcitabine arm.
Measure: Number; unit: participants
Arm/Group | Imexon + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 67 | 68
participants | 67 | 68

3. Secondary Outcome: Objective Response Rates of the Two Treatment Arms
Description: Objective response is measured by tumor reduction as defined in the RECIST criteria. Tumor shrinkage must be at least 30% to qualify as an objective response.
Time Frame: one year
Population: Per protocol, response evaluable population was treated and had baseline and at least one response evaluation.
Measure: Number; unit: percent of responses
Arm/Group | Amplimexon (Imexon) + Gemcitabine | Imexon Placebo + Gemcitabine
Number analyzed (Participants) | 53 | 55
percent of responses | 13.2 | 16.4

4. Secondary Outcome: Progression Free Survival
Description: To compare the median progression free survival (PFS) of the two treatment arms. Progression free survival is measured from randomization until the subject has documented disease progression by an objective measure. Subjects were censored if no documented progression had occurred at the one year time point. Subjects must be alive with no more than 20% increase in tumor size to qualify for progression free survival. Changes in tumor size are defined by RECIST criteria.
Time Frame: one year
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amplimexon (Imexon) + Gemcitabine | Imexon Placebo + Gemcitabine
Number analyzed (Participants) | 72 | 70
months | 2.8 [2.0 to 4.1] | 3.8 [2.2 to 4.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of treatment until the participant went off study treatment. This was an average timeframe of 4 months.
Description: Adverse event reporting was performed on the safety population. This included only those subjects that received at least one dose of drug. This was 67 subjects in the active arm and 68 in the placebo arm.
Arm/Group | Amplimexon (Imexon) + Gemcitabine | Imexon Placebo + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 51/67 | 44/68
Other Adverse Events (participants affected / at risk) | 66/67 | 68/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amplimexon (Imexon) + Gemcitabine (N=67) | Imexon Placebo + Gemcitabine (N=68)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hemoglobin (low) (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutrophils (low) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Conduction abnormality-AV block-third degree (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular arrhythmia-atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular arrhythmia-atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 7 (7) | 1 (1)
Death-death not otherwise specified (General disorders) | 0 (0) | 4 (4)
Death-disease progression not otherwise specified (General disorders) | 15 (15) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal (GI) other-gastrostromy (G) tube leak (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction-small bowel not otherwise specified (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stricture-biliary tree (Hepatobiliary disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Hemorrhage-abdomen not otherwise specified (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage-duodenum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage- lower gastrointestinal not otherwise specified (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage-nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhage-other gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage-upper gastrointestinal not otherwise specified (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatobiliary-other-biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver dysfunction (Hepatobiliary disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Fever-neutropenic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection with normal absolute neutrophil count-biliary tree (Infections and infestations) | 2 (3) | 1 (1)
Infection with normal absolute neutrophil count-blood (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal absolute neutrophil count-lung (pneumonia) (Infections and infestations) | 5 (5) | 4 (5)
Infection with normal absolute neutrophil count-cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Infection with unknown absolute neutrophil count-lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Edema:trunk/genital (General disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle weakness-whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Central nervous system ischemia (Nervous system disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 0 (0)
Pain-abdomen not otherwise specified (Gastrointestinal disorders) | 4 (4) | 4 (4)
Pain-back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain-chest/thorax not otherwise specified (General disorders) | 0 (0) | 2 (2)
Pain-pain not otherwise specified (General disorders) | 2 (2) | 0 (0)
Pain-stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 4 (4)
Renal-other-hemolytic uremic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Peripheral arterial ischemia (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 5 (5) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amplimexon (Imexon) + Gemcitabine (N=67) | Imexon Placebo + Gemcitabine (N=68)
Platelets (low) (Investigations) | 28 (100) | 32 (102)
Hemoglobin (low) (Blood and lymphatic system disorders) | 34 (84) | 36 (89)
Neutrophils (low) (Investigations) | 18 (55) | 32 (109)
Fatigue (General disorders) | 44 (75) | 44 (84)
Leukocytes (low) (Investigations) | 23 (84) | 17 (51)
Pain-abdomen not otherwise specified (Gastrointestinal disorders) | 33 (50) | 33 (61)
Nausea (Gastrointestinal disorders) | 42 (64) | 29 (44)
ALT (high) (Investigations) | 18 (49) | 16 (36)
Fever (General disorders) | 27 (49) | 18 (24)
AST (high) (Investigations) | 18 (38) | 14 (34)
Constipation (Gastrointestinal disorders) | 31 (41) | 26 (30)
Vomiting (Gastrointestinal disorders) | 25 (34) | 24 (37)
Edema:limb (General disorders) | 23 (31) | 27 (38)
Lymphopenia (Investigations) | 10 (35) | 11 (27)
Anorexia (Metabolism and nutrition disorders) | 23 (29) | 26 (30)
Diarrhea (Gastrointestinal disorders) | 21 (23) | 22 (36)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 (28) | 20 (29)
Alkaline phosphatase (high) (Investigations) | 13 (21) | 19 (31)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (18) | 13 (31)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (13) | 14 (26)
Hypokalemia (Metabolism and nutrition disorders) | 13 (18) | 11 (13)
Pain-extremity-limb (Musculoskeletal and connective tissue disorders) | 7 (12) | 11 (19)
Rash (Skin and subcutaneous tissue disorders) | 12 (18) | 10 (13)
Thrombosis/thrombus/embolism (Vascular disorders) | 12 (12) | 18 (19)
Rigors/chills (General disorders) | 16 (17) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The manuscript or abstract shall be submitted at least (45) days prior to submission for publication to permit Sponsor to request removal of any Confidential Information and to protect its rights to any patentable inventions set forth therein. Upon Sponsor's reasonable request, the investigator shall redact Sponsor's Confidential Information from any such proposed publication or shall delay publication for up to 90 days to permit Sponsor to protect its proprietary Information.